CLINICAL TRIAL: NCT05810181
Title: Gene Therapy Communication: Use of a Needs Assessment to Drive Decision-AIDS for Gene Therapy for Rare Diseases (GENETX)
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GENETX
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Young Adult: 15-25 parents/families of children (patients aged 8 and above) with rare genetic diseases, who have recently received gene therapy
  Interventions: Other: Interview
- Parent/caregiver: 10-20 patients/families of children with rare genetic diseases who were offered but have decided against receiving gene therapy or who were ultimately not eligible for a clinical trial.
  Interventions: Other: Interview
- Healthcare Worker: 10-20 health care workers' who provide care to patients receiving gene therapy.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — The following three groups of stakeholders will be interviewed to assess the beliefs, attitudes, and informational needs around gene therapy for rare pediatric diseases:
  (1) patients and families of children with rare genetic diseases who have received gene therapy (to assess their perspectives and understand their informational needs around participating in a clinical trial using gene therapy), (2) patients and families of children with rare genetic diseases who were offered but have decided against receiving gene therapy or ultimately did not qualify for a trial (to elicit feedback and to evaluate whether their informational needs and communication expectations about participating in a clinical trial using gene therapy were met), and (3) healthcare workers who provide care to patients receiving gene therapy (to assess their perspective regarding patient/family needs for gene therapy education and communication).

SUMMARY:
This prospective mixed-method interview study aims to qualitatively describe the beliefs, attitudes, and informational needs around gene therapy for rare pediatric diseases among patients and parents of children with a rare disease targeted for treatment using gene therapy techniques. Using learned insights, the team will develop an online platform providing educational content and patient decision aids for patients and their families.

DETAILED DESCRIPTION:
The study team seeks to understand the unique needs of patients and parents of children who are considering novel experimental gene therapy treatments. The study team will engage patient, caregiver, and healthcare worker stakeholders to understand their attitudes, beliefs, and concerns surrounding these treatments. Based on these insights, the team, with the support of the above stakeholders and an external vendor, will develop web platform offering educational content and decision aids to enhance their experience and overall satisfaction with the process of making treatment decisions. This is especially important as novel therapies for SCD will increasingly include gene editing in pediatric trials over the next two years. These efforts will address significant gaps in the educational material available to those considering gene therapy and (to the team's knowledge) will create a resource that will be the first of its kind.

ELIGIBILITY:
Inclusion Criteria:

1. For Group 1 participants only (Undergone Gene Therapy):

   * Parent/caregiver whose child has undergone gene therapy. OR Parent/caregiver of a child who died after receiving gene therapy at least 6 months prior to enrollment, but no more than 24 months prior to enrollment, to be contacted no sooner than 3 months after the death has occurred and no longer than 2 years. OR Patients age 8 and above who have undergone gene therapy.
   * Willingness to participate in one-on-one video interview with a study team member using a personal mobile device or computer with working internet connection.
   * Must be willing to provide verbal informed consent.
   * Release of information form signed by participant providing our study team with permission to contact healthcare provider to verify their diagnosis and receipt of gene therapy (if received).
   * Successful verification of diagnosis of rare genetic disease targeted for treatment using gene therapy.
   * A positive confirmation on receipt of gene therapy and type received from their healthcare provider (only for those received gene therapy).
2. For Group 2 participants only (Offered, but did not Undergo Gene Therapy):

   * Parent/caregiver of children (or patients 8 and above ) with a rare genetic disease who had been offered but were not eligible for a trial or decided against receiving gene therapy.
   * Willingness to participate in one-on-one video interview with a study team member using a personal mobile device or computer with working internet connection.
   * Must be willing to provide verbal informed consent.
   * Signed release of information form providing GeneTx study team with permission to contact participant's healthcare provider to verify the diagnosis.
   * Successful verification of diagnosis of rare genetic disease targeted for treatment using gene therapy.
3. For Group 3 participants only (Provider Interviews):

   * Healthcare worker who has provided care to ≥ 2 patients receiving gene therapy.
   * Willingness to participate in one-on-one video (or in-person) interview with a study team member using a personal mobile device or computer with working internet connection.
   * Informed consent from a study participant.

Exclusion Criteria:

* Participants who are unable to converse fluently in English will be excluded.
* Inability or unwillingness of research participant to give verbal informed consent.
* Participants who lack access to a computer or mobile device that supports video communications will be excluded.
* Condition or chronic illness, which in the opinion of the PI/Co-I, makes participation unsafe or untenable (i.e., cognitive impairment, concurrent acute morbidity).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: About 45-50 patients (age 8 and above) or parents of children verified to have a rare disease targeted for treatment using gene therapy techniques and 10-20 healthcare workers who provide care to patients receiving gene therapy.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Use of semi-structured interviews to assess the beliefs, attitudes, and informational needs around gene therapy among patients and families with rare genetic diseases. | 2 years
  Trained experts will interview study participants to elucidate their beliefs, attitudes, and informational needs around gene therapy for rare pediatric diseases among the disease stakeholders. These interviews will be analyzed via the well-described rigorous methodology of semantic content analysis to identify themes through a systematic and standardized process.

CONTACTS AND LOCATIONS:
Overall Officials: Liza-Marie Johnson, MD, MPH, MSB, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States